CLINICAL TRIAL: NCT01803165
Title: Lower Extremity Regional Anesthesia and Infrainguinal Bypass Grafting
Status: Withdrawn | Type: Observational
Why Stopped: Inadequate patient population
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0541-12-EP
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Vascular Disease
Keywords: emesis,post operative.; cognitive dysfunction, post operative.; wound infection, post operative.; pain, post operative.; Anesthesia, Conduction/methods; Anesthesiology/methods; Arteriovenous Shunt, Surgical/adverse effects; Regional Blood Flow/drug effects; Risk Factors; Thrombosis; Treatment Outcome; Vascular Surgical Procedures/methods; Vasodilation/drug effects
MeSH Terms: conditions — Peripheral Vascular Diseases; Cognitive Dysfunction; Wound Infection; Pain, Postoperative; Arteriovenous Fistula; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Single shot femoral and sciatic nerve block: Prospective patient study group who present for infrainguinal bypass grafting and will receive single shot femoral and sub gluteal sciatic nerve blocks.
  Interventions: Procedure: Single shot femoral and sciatic nerve block
- Retrospective study group: Retrospective chart review will be performed and data collected on patients who have undergone infrainguinal bypass grafting under general anesthesia and without the use of regional or neuraxial anesthesia.

INTERVENTIONS:
Procedure: Single shot femoral and sciatic nerve block — Ultrasound will be performed with a linear 10- to 13-Megahertz probe while performing the nerve block. Standard American Society of Anesthesiology monitors will be applied and the patient sedated at the discretion of the anesthetic team. Complications such as vascular puncture, pain on injection, or systemic toxicity will be recorded. A perineural dosing regimen for the regional blocks will be as follows: (femoral block) 20cc of 0.5% ropivicaine and (sub-gluteal posterior sciatic block) 20cc of 0.2% ropivicaine. Epinephrine will be withheld from the local anesthetic in order to prevent the potential of further ischemic complications.
  Groups: Single shot femoral and sciatic nerve block

SUMMARY:
In this investigation, the investigators will attempt to demonstrate that patients who have received nerve blocks (regional anesthesia) prior to open surgical vascular bypass of the lower extremities (infrainguinal bypass grafting) will have improved surgical outcomes namely a reduction in the rates of death, wound infection, graft thrombosis, graft revision, and amputation. As well, the investigators anticipate that patients who have undergone regional anesthesia for infrainguinal bypass grafting will have improved secondary outcomes with respect to a decreased length of stay, narcotic consumption, nausea and vomiting, post-operative cognitive dysfunction, major cardiac events, post-operative pain, and hyperglycemic episodes.

DETAILED DESCRIPTION:
Background The post-operative benefits of regional anesthesia have been described in patients undergoing vascular access surgery(1, 2). Some of the benefits that have been identified are improved vascular flow, decreased thrombosis rates, and early maturation of grafts(2). It is speculated that these benefits can be mainly attributed to sympathetic blockade by regional anesthesia. Recent literature review has not identified any prior studies which have attempted to prospectively identify if there are improved surgical outcomes in patients undergoing revascularization surgery when regional anesthesia is utilized. However, Kashyap et al. reported that regional anesthesia may decrease the incidence of perioperative thrombosis in patients who had undergone infra-popliteal revascularization surgery over a 20 year period(3). In this investigation we will attempt to ascertain whether or not there will be improved surgical outcomes namely a reduction in the rates of death, wound infection, graft thrombosis, graft revision, and amputation. As well, we anticipate that patients who have undergone regional anesthesia for infrainguinal bypass grafting will have improved secondary outcomes with respect to a decreased length of stay, narcotic consumption, nausea and vomiting, post-operative cognitive dysfunction, major cardiac events, post-operative pain, and hyperglycemic episodes.

Methods After Investigational Review Board approval, written informed consent will be obtained from 20 patients undergoing fem-popliteal bypass surgery at University of Nebraska Medical Center and enrolled in our prospective cohort registry. Patients will be excluded from the study if age is less than 19 years, allergies to amide anesthetics, inability to undergo general anesthesia, acute limb ischemia, any existence of contraindications to regional anesthesia in the presence of antiplatelet or anticoagulative drugs, or evidence of gross neurological dysfunction of the lower extremity. Baseline health data of the patient will be recorded. Ultrasound will be performed with a linear 10- to 13-Megahertz probe while performing the nerve block. Standard American Society of Anesthesiology monitors will be applied and the patient sedated at the discretion of the anesthetic team. Complications such as vascular puncture, pain on injection, or systemic toxicity will be recorded. A perineural dosing regimen for the regional blocks will be as follows: (femoral block) 20cc of 0.5% ropivicaine and (sub-gluteal posterior sciatic block) 20cc of 0.2% ropivicaine. Epinephrine will be withheld from the local anesthetic in order to prevent the potential of further ischemic complications. The patient will then undergo general anesthesia at the discretion of the anesthetic team. Any anesthetic or surgical complication will be recorded during the OR interval. The type of graft utilized and specific location of arterial intervention will be recorded.

Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital. Primary outcomes which will be recorded include: death, wound infection, graft thrombosis, graft revision, and amputation. Secondary outcomes which will be recorded are pain scores, nausea and vomiting, 24 hour narcotic consumption, graft failure (defined as any occlusion requiring return to operating room), any related return to the OR for the index procedure, any major adverse cardiac events (MACE), administration of warfarin or antiplatelet medications, average 24 hour blood sugar, creatinine levels, postoperative cognitive dysfunction, and requirement of supplemental oxygen upon discharge from the PACU. As well, the patient will be queried for resumption of tobacco products. The patient's length of hospital stay will be recorded.

On discharge there will be continued surveillance for the following primary outcomes: death, wound infection, graft thrombosis, graft revision, and amputation. The secondary outcomes which will be recorded are as follows: presence of pain at rest, pain on ambulation, continued administration of anticoagulants or antiplatelets, graft failure (defined as any occlusion requiring return to operating room), any related return to the OR for the index procedure, any major adverse cardiac events (MACE), average 24 hour blood sugar, creatinine levels, and all ankle brachial pressure index (ABPI) and doppler ultrasound reports will be recorded. Also, patients will be queried for resumption of tobacco products. These observations will be recorded on post-operative day 7, 31, and 93.

A comparison group of patients (N=20) who have undergone infra-inguinal bypass grafting will be obtained from retrospective chart review. Patients who have undergone regional or neuroaxial anesthesia for their bypass procedure will be excluded. As well, patients will be matched to their cohorts by age, sex, health comorbidities including: Congestive heart failure, smoking, diabetes, and renal dysfunction, and chronic anticoagulants or antiplatelet medication administration. The same primary and secondary outcome data obtained in the prospective portion of this study will be sought and recorded by chart review.

Conclusion Improved vascular surgical outcomes have been described in patients receiving regional anesthesia and neuroaxial anesthesia(2-4). Specifically, we anticipate a decrease in overall rates of death, wound infection, graft thrombosis, graft revision, and amputation in patients receiving regional anesthesia for infra-inguinal bypass grafting. As well, we hypothesize that patients receiving regional anesthestics will have improved secondary outcomes including decreased length of stay, narcotic consumption, nausea and vomiting, post-operative cognitive dysfunction, cardiac events, post-operative pain, and hyperglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years of age and older who are candidates to undergo infrainguinal bypass grafting for the treatment of peripheral vascular disease

Exclusion Criteria:

* age is less than 19 years
* allergies to amide anesthetics
* inability to undergo general anesthesia
* acute limb ischemia
* any existence of contraindications to regional anesthesia in the presence of antiplatelet or anticoagulative drugs
* evidence of gross neurological dysfunction of the lower extremity

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 19 years of age and older who are candidates to undergo infrainguinal bypass grafting for the treatment of peripheral vascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Estimated); Primary Completion 2013-09-10 (Actual); Study Completion 2013-09-10 (Actual)

PRIMARY OUTCOMES:
graft thrombosis | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for thrombosis, the predominant mechanism of early graft failure. This continues post-discharge.
limb amputation | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for the need for limb amputation. This continues post-discharge.
wound infection | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for wound infection. This continues post-discharge.
graft revision | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for the need for graft revision. This continues post-discharge.
death rate | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for expiration. This continues post-discharge.

SECONDARY OUTCOMES:
decreased length of hospital stay | up to 1 month
  decreased length of post surgical hospital stay
narcotic consumption | up to 3 months
  Overall narcotic consumption will be recorded
nausea and vomiting | up to 1 month
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for nausea and vomiting. This continues post-discharge.
post-operative cognitive dysfunction | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for cognitive dysfunction. This continues post-discharge.
major cardiac events | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for major cardiac events. This continues post-discharge.
post-operative pain | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for post-operative pain. This continues post-discharge.
hyperglycemic episodes | up to 3 months
  Following surgery, the patient will be monitored and data recorded daily while the patient is recovering in the hospital for hyperglycemic episodes. This continues post-discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Nicholas, MD, Principal Investigator — Univversity of Nebraska Medical Center

REFERENCES:
- [Background] Malinzak EB, Gan TJ. Regional anesthesia for vascular access surgery. Anesth Analg. 2009 Sep;109(3):976-80. doi: 10.1213/ane.0b013e3181adc208. PMID 19690276
- [Background] Sahin L, Gul R, Mizrak A, Deniz H, Sahin M, Koruk S, Cesur M, Goksu S. Ultrasound-guided infraclavicular brachial plexus block enhances postoperative blood flow in arteriovenous fistulas. J Vasc Surg. 2011 Sep;54(3):749-53. doi: 10.1016/j.jvs.2010.12.045. Epub 2011 Mar 2. PMID 21367563
- [Background] Kashyap VS, Ahn SS, Quinones-Baldrich WJ, Choi BU, Dorey F, Reil TD, Freischlag JA, Moore WS. Infrapopliteal-lower extremity revascularization with prosthetic conduit: a 20-year experience. Vasc Endovascular Surg. 2002 Jul-Aug;36(4):255-62. doi: 10.1177/153857440203600402. PMID 15599475
- [Background] Singh N, Sidawy AN, Dezee K, Neville RF, Weiswasser J, Arora S, Aidinian G, Abularrage C, Adams E, Khuri S, Henderson WG. The effects of the type of anesthesia on outcomes of lower extremity infrainguinal bypass. J Vasc Surg. 2006 Nov;44(5):964-8; discussion 968-70. doi: 10.1016/j.jvs.2006.06.035. Epub 2006 Sep 26. PMID 17000075